CLINICAL TRIAL: NCT02206321
Title: Comparison of Navigation and Conventional Total Knee Arthroplasties
Brief Title: Effects of Computer Navigation Versus Conventional Total Knee Arthroplasty on Endothelial Damage Marker Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jih-Yang Ko, Professor, Chang Gung Memorial Hospital
Other Study IDs: IRB 100-0038A3; ChangGungMH (Other: ChangGungMH)
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Computer-assisted Navigation Versus Conventional Total Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Obtain the serum and hemovac drainage from the patients, and analyze the concentrations of the markers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Navigation total knee arthroplasty: Navigation total knee arthroplasty
  Interventions: Procedure: Navigation total knee arthroplasty
- Conventional total knee arthroplasty: Conventional total knee arthroplasty
  Interventions: Procedure: Conventional total knee arthroplasty

INTERVENTIONS:
Procedure: Navigation total knee arthroplasty — computer assisted navigation total knee arthroplasty without femur intramedullary involvement
  Groups: Navigation total knee arthroplasty
Procedure: Conventional total knee arthroplasty — conventional technique with femur intramedullary violation
  Groups: Conventional total knee arthroplasty

SUMMARY:
1. Prospective follow-up and comparative analysis of early, midterm, and long-term surgical results and complications between navigation assisted TKA and conventional TKA.
2. Prospective comparative analysis of cytokines (including ICAM, VCAM, and PECAM) from blood, tissues, and drainage between navigation assisted TKA and conventional TKA.
3. Prospective follow-up of surgical results of navigation-assisted TKA.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most successful surgery in orthopaedic field. However, occasional outliner from perfect alignment after prosthesis implantation and unavoidable complications are still concerns. The usage of navigation-assisted system on total knee arthroplasty has provided better accuracy of the component alignment and quantity in knee kinematics, which theoretically affords better and consistent functional outcome.

In addition to better alignment, the design of navigation system avoids violation of the medullary canal. This less invasive environment might be contributable to the less blood loss in the drainage bottle, less blood transfusion more stable hemodynamic status, fewer hospitalization days, and fewer complications.

Systemic emboli phenomena during preparation of the femur and tibia are well recognized during total knee arthroplasty. They are widely believed to be the cause of intraoperative hypotension and reduced cardiac output, which may lead to circulatory collapse, change of mental status or cerebral infarction. Kalairajah et al reported that navigation-assisted total knee arthroplasty, when compared with conventional jig-based surgery, significantly reduces systemic emboli as detected by transcranial Doppler ultrasonography. Church et al undertook a prospective, double-blind, randomized study to compare the cardiac emboli load by tranesophageal echocardiography and demonstrated that computer-assisted TKA resulted in the release of significant fewer systemic emboli than the conventional procedure using intramedullary alignment. The increased blood loss in conventional TKA may be due to intramedullary jigging of both femur and tibia, bleeding from sinusoids at the cut cancellous bone surfaces with continuous suction drainage and more soft tissue dissection during balancing of the prosthesis. The investigators have underwent more than 730 computer-assisted TKA since 2005. The investigators data shows less bleeding and fewer transfusion after navigation assisted TKA. The investigators wish to further follow-up and delineate the differential clinical outcomes and perioperative markers (including ICAM, VCAM, and PECAM and other cytokines )between computer-assisted TKA and conventional TKA.

ELIGIBILITY:
Inclusion Criteria:

* degenerative osteoarthritis of the knee

Exclusion Criteria:

* autoimmune diseases, rheumatoid arthritis, malignancies, previous knee surgery or post-traumatic arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients were recruited from the patient undergoing scheduled total knee arthroplasty in our hospitals (Chang Gung Memorial Hospital, Kaohsiung medical center).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
ELISA analysis to compare concentrations of target molecules in serum and hemovac drainage between two groups | 24 hours after surgery
  We collect the serum and sample from hemovac drainage 24 hours after the surgery, to measure the concentrations of target molecules (ICAM, VCAM, PECAM).

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Yang Ko, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Kuo SJ, Wang FS, Wang CJ, Ko JY, Chen SH, Siu KK. Effects of Computer Navigation versus Conventional Total Knee Arthroplasty on Endothelial Damage Marker Levels: A Prospective Comparative Study. PLoS One. 2015 May 8;10(5):e0126663. doi: 10.1371/journal.pone.0126663. eCollection 2015. PMID 25955252